CLINICAL TRIAL: NCT03332537
Title: Precision Pain Self-Management in Young Adults With Irritable Bowel Syndrome
Acronym: IBS-SM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Xiaomei Cong, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H16-152; 1P20NR016605-01 (NIH)
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Young Adults; IBS; Self Management; Pain; Gut microbiome; Genetics; Online education
MeSH Terms: conditions — Irritable Bowel Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Using a stratified and blocked randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will be provided an online interactive platform to access electronic modules (total of 10) on: IBS-related pain neurophysiology and the brain-gut axis and self-management strategies. There is no additional intervention.
- Personalized IBS Pain SM (Experimental): Participants will be enrolled in the online platform. After completion of the modules, they will be scheduled for a consultation with a research nurse about their level of peripheral and central sensitivity, self-evaluation of IBS-pain SM, goal setting and self-monitoring of IBS-pain and physical activity. They will be asked to document their pain and all symptom SM behaviors daily for the next 10 weeks. At the 6-week follow-up visit, the researcher will review the online activities of the participant, go over the previously selected goals with the participants. The study nurse will acknowledge accomplishment of goals and assist in problem-identification and solving.
  Interventions: Behavioral: Personalized IBS Pain SM

INTERVENTIONS:
Behavioral: Personalized IBS Pain SM
  Arms: Personalized IBS Pain SM

SUMMARY:
This pilot project will provide foundational information about the contextual factors of irritable bowel syndrome (IBS) related pain (pain catastrophizing, perceived stress, reactivity pain sensitivity, genetic and microbiome) on pain self-management (SM) process and outcomes. In addition, the investigators will gain insight on the potential impact of the personalized IBS-pain SM approach on pain SM behaviors and health outcomes.

DETAILED DESCRIPTION:
Intense, recurrent abdominal (visceral) pain is a predominant symptom of irritable bowel syndrome (IBS), a functional gut disorder that typically manifests in the early adult years. IBS is common with prevalence reaching over 20% in some regions of the world, and affects more women than men. While women report more severe IBS-related pain, both younger men and women report more severe pain compared to older adult cohorts. Direct costs of care and lost productivity in the U.S. exceed $21 billion annually, and individuals with IBS utilize more healthcare services than the general population, including outpatient visits, diagnostic testing and over-the-counter and prescription medications. Individuals with IBS report that pain is the most distressing symptom and has the greatest impact on quality of life, however, current approaches to improve self- management of IBS-related pain do not target individual, context-specific factors of pain. Therefore, individuals with IBS-related pain often endure a long and frustrating course of learning how to manage pain on their own accord. The proposed pilot project was developed based on this common situation and will provide feasibility data about the influence of providing a personalized pain SM intervention to individuals with IBS-related pain. IBS-related pain is associated with sensitization of the central nervous system, and approximately half of all patients with IBS have visceral hypersensitivity. These alterations in pain processing escalate pain perception, and can increase vulnerability to other co-morbid pain disorders which individuals with IBS frequently suffer. Pain sensitization is influenced by pain-sensitivity genes and, specific to IBS-related pain, the gut microbiome. Therefore, as contextual factors of pain associated with IBS, the investigators will measure peripheral and central sensitivity, single-nucleotide polymorphisms (SNPs) of candidate pain-sensitivity genes and the gut microbiome. The SM intervention was designed to provide factual information about IBS pain, triggers of pain and pain SM skills. The experimental group will receive one-on-one consultation tailored around the individual's assessment results of peripheral and central pain sensitivity as measured by quantitative sensory testing (QST) and targeted toward increasing pain self-efficacy and self-regulation skills and abilities. The proposed pilot project will provide foundational information about the contextual factors of IBS pain (pain catastrophizing, perceived stress, reactivity pain sensitivity, genetic and microbiome) on pain SM process and outcomes. In addition, the investigators will gain insight on the potential impact of the personalized IBS-pain SM approach on pain SM behaviors and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-29 years of age
* Diagnosis of IBS from a healthcare provider with a current report of pain
* Able to read and write in English
* Daily access to a computer connected to the internet

Exclusion Criteria:

* Other chronic painful conditions (i.e. fibromyalgia, chronic pelvic pain, or chronic interstitial cystitis)
* Infectious disease (hepatitis, HIV, MRSA)
* Celiac disease or inflammatory bowel disease
* Diabetes Mellitus
* Serious mental health conditions (ex. Bipolar disorder, schizophrenia, mania)
* Women who are pregnant or post-partum in last 3 months
* Regular use of opioids, iron supplements, prebiotics/probiotics or antibiotics, or substance abuse.
* Injury to non-dominant hand or presence of open skin lesions

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pain sensitivity | Baseline and 6 weeks and 12 weeks
  Quantitative sensory testing - Change over time
Change in gut microbiome | Baseline and 6 weeks and 12 weeks
  Change over time

SECONDARY OUTCOMES:
Genetic variations (Pain-susceptibility SNPs genotyping) | Baseline
  related to IBS-related pain and gut microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Cong, PhD, RN, Principal Investigator — University of Connecticut
Locations (2):
- United States (2):
  - UConn Health Center, Farmington, Connecticut
  - University of Connecticut, Storrs, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that are part of National Institute of Nursing Research (NINR) designated common data elements collected during the trial, after de-identification have been submitted to NIH repository at the Common Data Repository for Nursing Science (cdRNS). Data can be accessed by directly submitting requests at that website.
  When will data be available (start and end dates)? Immediately. No end date.
  With whom? Anyone who wishes to access the data and creates an account on cdRNS.nih.gov.
  By what mechanism will data be made available? Data are available at cdRNS.nih.gov
Time Frame: within 2 years
Access Criteria: Requests will be submitted through the cdRNS website
URL: https://cdrns.nih.gov/access-data

REFERENCES:
- [Derived] Chen J, Zhang Y, Barandouzi ZA, Lee J, Zhao T, Xu W, Chen MH, Feng B, Starkweather A, Cong X. The effect of self-management online modules plus nurse-led support on pain and quality of life among young adults with irritable bowel syndrome: A randomized controlled trial. Int J Nurs Stud. 2022 Aug;132:104278. doi: 10.1016/j.ijnurstu.2022.104278. Epub 2022 Apr 30. PMID 35640500